CLINICAL TRIAL: NCT06831058
Title: A Pilot Study of Efgartigimod for Immune-mediated Thrombotic Thrombocytopenic Purpura (iTTP)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOT-2024-32825
Record Dates: First submitted 2025-02-13; First posted 2025-02-17 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Immune-mediated Thrombotic Thrombocytopenic Purpura
MeSH Terms: interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- iTTP patients (Experimental): participants with a history of iTTP in clinical remission but with ADAMTS13 deficiency (>30% but < 70% activity)
  Interventions: Drug: efgartigimod

INTERVENTIONS:
Drug: efgartigimod — intravenous efgartigimod weekly with monitoring of ADAMTS13 activity for 8 weeks, followed by an observational period of 8 weeks or until treatment failure.

SUMMARY:
Immune-mediated Thrombotic thrombocytopenic purpura (iTTP) is a rare, autoimmune disorder characterized by life-threatening episodes of thrombocytopenia, microangiopathic hemolytic anemia and organ damage. Patients have an unpredictable course punctuated by relapses associated with autoantibody-mediated (primarily IgG) depletion of ADAMTS13, a key regulator of coagulation. ADAMTS13 deficiency during remission has been associated with increased risk of relapse, but also, and potentially more devastating, ischemic stroke.

Until recently, it was presumed that rituximab (a monoclonal antibody targeting B cells) improved relapse-free survival in most patients, but this was based on findings from very small studies. Given concern about stroke and relapse risk, preventive immunosuppression with rituximab has also recently come into practice for patients with falling ADAMTS13 activity (ADAMTS13-relapse). It is expected that following efgartigimod therapy, there will be a rise in ADAMTS13 activity to the normal range that will be sustained during the treatment period. Following withdrawal of therapy, it is expected that most participants will experience a fall in ADAMTS13 activity, demonstrating the safety and efficacy in efgartigimod to reliably but temporarily reduce pathogenic antibodies. This would demonstrate the potential efficacy for efgartigimod as a maintenance therapy to safely prevent relapse of iTTP to be further explored in a larger efficacy study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide a signed informed consent form
2. Subject is 18 years or older at the time of screening
3. Subject has a prior history of iTTP as defined by the presence of ADAMTS13 activity < 10% with ADAMTS13 antibodies or inhibitor, thrombocytopenia (platelet count < 100) and microangiopathic hemolytic anemia (defined by the presence of schistocytes on blood smear)
4. Subject is in clinical remission from iTTP (normal platelet count) for at least 90 days
5. Subject has ADAMTS13 activity < 70% and > 30% on 2 separate occasions separate by at least 7 days
6. Subject is at least 6 months from last dose of rituximab or other intravenous immunosuppression
7. If taking other oral immunosuppressants, no change in dose for at least 60 days
8. Female subjects of childbearing potential must present with a negative pregnancy test and agree to employ highly effective birth control measures for duration of study.

Sexually active male subjects must agree to use an effective method of contraception for the duration of the study

Exclusion Criteria:

1. Subject has been diagnosed with cTTP
2. Subject has been exposed to another investigational product within 30 days prior to enrollment or is scheduled to participate in another clinical study involving investigational product or investigational device during the course of the study
3. Subject is unable to understand the nature, scope, and possible consequences of the study.
4. Subject is pregnant or lactating
5. Subject has a known life-threatening hypersensitivity reaction to efgartigimod

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
safety of efgartigimod by the incidence of relapse | 8 weeks post-intervention
  Relapse rate in the experimental arm compared with the historical rituximab arm
safety and tolerability of efgartigimodhistorical rituximab arm | 8 weeks post-intervention
  Incidence and severity of adverse events (AEs), AEs of special interest (AESIs) and serious AEs (SEAs)
efficacy of efgartigimod to achieve a normal ADAMTS13 activity by Day 60 of the study | 60 days
  Compare the mean ADAMTS13 activity and proportion with normal ADAMTS13 activity at Day 60 and 90 between the experimental and historical cohorts
efficacy of efgartigimod to prevent the need for other preemptive therapy to rescue severe ADAMTS13 deficiency | 8 weeks post-intervention
  Compare the rate use of rescue therapy between the experimental and historical cohort treated with preemptive rituximab, as required by the lack of ADAMTS13 activity increase by 20%

SECONDARY OUTCOMES:
the efficacy of efgartigimod to raise ADAMTS13 activity more rapidly than historically treated patients with rituximab | Day 60 and day 90
  Compare the mean slope of ADAMTS13 rise at the end of treatment (Day 60) and at 90 days between cohorts
the efficacy of efgartigimod to deplete pathogenic ADAMTS13 antibodies | 8 weeks post-intervention
  Compare the mean ADAMTS13 antibody titers and proportion with >50% reduction in antibody titer between cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Mazepa, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No